CLINICAL TRIAL: NCT05219578
Title: A Phase 1/2 Study of RTX-224 for the Treatment of Patients With Advanced Solid Tumors
Brief Title: RTX-224 Monotherapy in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor terminated study after dosing 2 dose groups (7 pts) and closed trial on 11/30/22. RTX-224 was well-tolerated with no DLTs, no related deaths, SAEs or Gr. 3/4 AEs and cleared rapidly (w/in 10 min).
Sponsor: Rubius Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTX-224-01
Record Dates: First submitted 2022-01-06; First posted 2022-02-02 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Non Small Cell Lung Cancer; Cutaneous Melanoma; Head and Neck Squamous Cell Carcinoma; Urothelial Carcinoma; TNBC - Triple-Negative Breast Cancer
Keywords: Solid Tumor, Advanced Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RTX-224 Dose Escalation (Experimental): Phase 1: RTX-224 monotherapy dose escalation in Solid Tumors, administered intravenously on Day 1 of each cycle.
  Interventions: Drug: RTX-224
- RTX-224 Dose Expansion (Experimental): Phase 2: RTX-224 monotherapy dose expansion in Solid Tumors, administered intravenously on Day 1 of each cycle.
  Interventions: Drug: RTX-224

INTERVENTIONS:
Drug: RTX-224 — RTX-224 monotherapy

SUMMARY:
This is an open-label, multidose, first-in-human (FIH), Phase 1/2 study of RTX-224 for the treatment of patients with relapsed or refractory (R/R), or locally advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open label, multicenter, multidose, first-in-human (FIH), dose escalation and expansion to determine the safety and tolerability, recommended phase 2 dose, and pharmacology, and antitumor activity of RTX-224 in adult patients with persistent, recurrent, or metastatic, unresectable solid tumors. The study will include a monotherapy dose escalation phase followed by an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures Patients ≥18 years with an ECOG of 0 or 1
* R/R, or locally advanced, unresectable, and histologically or cytologically confirmed

  (a) NSCLC, (b) cutaneous melanoma, (c) HNSCC, (d) UC, or (e) TNBC, which are refractory to or otherwise ineligible for treatment with standard-of-care treatments
* Prior therapy in each disease setting must include the following:

  * NSCLC: Patients must have experienced disease progression following platinum-containing chemotherapy and a PD-1 or PD-L1 inhibitor. Patients with EGFR, ALK, ROS-1, or other actionable mutations should have previously received or been ineligible for therapies targeting their respective mutation(s).
  * Cutaneous melanoma: Patients must have experienced disease progression following a PD-1 or PD-L1 inhibitor. Patients with V600E mutations should have previously received or been ineligible for approved BRAF inhibitor or MEK inhibitor therapy.
  * HNSCC: Patients must have experienced disease progression following platinum-based combination chemotherapy and a PD-1 or PD-L1 inhibitor.
  * UC: Patients must have experienced disease progression following platinum-based combination chemotherapy and a PD-1 or PD-L1 inhibitor.
  * TNBC: Patients must have experienced disease progression following single-agent or combination chemotherapy. Patients with BRCA1/2 mutations should have previously received or been ineligible for an approved PARP inhibitor; patients who are PD-L1 positive should have received or been ineligible for an approved PD-1 or PD-L1 inhibitor.
* Disease must be measurable per Response Evaluation Criteria
* The shorter of 28 days or 5 half-lives must have elapsed since the completion of prior therapy, before initiation of study treatment.
* Adequate Organ Function as Defined by the protocol:

  * AST and ALT ≤3 × the upper limit of normal (ULN) Except in documented cases of Gilbert syndrome, total bilirubin ≤1.5 × ULN
  * Serum albumin ≥2.5 g/dL
  * Serum or plasma creatinine ≤1.5 × ULN and/or glomerular filtration rate ≥50 mL/min/1.73 calculated by the Cockcroft-Gault formula
  * Absolute neutrophil count ≥1 × 103/μL
  * Platelet count ≥100 × 103/μL
  * Hemoglobin ≥9 g/dL

Exclusion Criteria:

* Patient has central nervous system (CNS) involvement. If the patient fulfills the following 3 criteria, she/he is eligible for the trial after consultation with the Sponsor Medical Monitor.
* Completed prior therapy for CNS metastases (radiation and/or surgery)
* CNS tumor(s) is clinically stable at the time of enrollment
* Patient does not require corticosteroid or antiepileptic therapy for management of CNS metastases
* Known hypersensitivity to any component of study treatment or excipients.
* Positive antibody screen using institution's standard type and screen test.
* Clinically significant, active and uncontrolled infection, including human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Safety Assessment by rate of Adverse Events (AEs) | up to 30 months
  Measured by incidence of Treatment Emergent Adverse Events (TEAEs)
Dose limiting toxicities (DLTs) of RTX-224 | up to 30 months
  As determined by incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacodynamics (PD) of RTX-224 | up to 30 months
  As measured by the changes in immune cell populations, e.g., T cells and NK cells
Pharmacokinetics (PK) of RTX-224 | up to 30 months
  Maximum concentration (Cmax) of RTX-224 cells (positive for both 4-1BBL and IL-12 using flow cytometry) in blood after administration will be measured.
Pharmacokinetics (PK) of RTX-224 | up to 30 months
  Time to maximum concentration (tmax) of RTX-224 cells (positive for both 4-1BBL and IL-12 using flow cytometry) in blood after administration will be measured.
Anti-tumor activity of RTX-224 | up to 30 months
  As measured by duration of response (DoR)
Anti-tumor activity of RTX-224 | up to 30 months
  As measured by overall survival (OS)
Anti-tumor activity of RTX-224 | up to 30 months
  As measured by progression free survival (PFS)
Anti-tumor activity of RTX-224 | up to 30 months
  As measured by disease control rate (DCR)
Anti-tumor activity of RTX-224 | up to 30 months
  As measured by objective response rate (ORR)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth, Scottsdale, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco Health, San Francisco, California
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No